CLINICAL TRIAL: NCT06016894
Title: Comparative Study Between Hydroxyapetite Nanoparticles and Tricalcium Phosphate Nanoparticles Loaded on Platelet Rich Fibrin Membranes for Treatment of Gingival Recession
Brief Title: Hydroxyapetite Nanoparticles, Tricalcium Phosphate Nanoparticles, and PRF for Treatment of Gingival Recession
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Enas Elgendy, Prof. of Oral Medicine and Periodontology, October 6 University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: khafrelsheikh university
Record Dates: First submitted 2023-08-24; First posted 2023-08-30 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis | interventions — Prolactin-Releasing Hormone

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nanocrystalline hydroxyapatite (Active Comparator): Nanocrystalline hydroxyapatite loaded in PRF+ coronally advanced flap
  Interventions: Procedure: coronally advanced flap; Other: Nanocrystalline hydroxyapatite loaded in PRF
- Nanocrystalline tricalcium phosphate (NcTCP) (Active Comparator): Nanocrystalline tricalcium phosphate (NcTCP) loaded in PRF+ coronally advanced flap
  Interventions: Procedure: coronally advanced flap; Other: Nanocrystalline tricalcium phosphate loaded in PRF

INTERVENTIONS:
Procedure: coronally advanced flap — coronally advanced flap operation
Other: Nanocrystalline hydroxyapatite loaded in PRF — Nanocrystalline hydroxyapatite loaded in PRF
  Arms: Nanocrystalline hydroxyapatite
Other: Nanocrystalline tricalcium phosphate loaded in PRF — Nanocrystalline tricalcium phosphate (NcTCP) loaded in PRF
  Arms: Nanocrystalline tricalcium phosphate (NcTCP)

SUMMARY:
The aim of the present study was to compare between nanocrystalline hydroxyapatite and tricalcium phosphate carried on PRP membrane in treatment of Miller's class 1 gingival recession in human.

DETAILED DESCRIPTION:
gingival recession (GR) is apical movement of the gingival margin beyond the cement-enamel junction. The use of free gingival grafts, sliding pedicle grafts, subepithelial connective tissue grafts, envelope or tunnelling techniques, the use of acellular dermal, connective tissue allografts, guided tissue regeneration, Platelet rich fibrin (PRF), and coronally advanced flap (CAF) are the surgical methods that have been developed to treat gingival recession. For treatments of intrabony defects, a synthetic nanocrystalline hydroxyapatite (NcHA) bone graft has been introduced. Osteoconductivity, bioresorbability, and close contact are benefits of NcHA material. Critical size defects showed quick healing when the NcHA was utilised as a bone graft alternative. NcHA binds to bone and increases osteoblast activity to promote bone regeneration. A promising bone replacement material, tricalcium phosphate (TCP) is known for its strong bioactivity and resorbable qualities. Tricalcium phosphate (TCP) is one of the most popular and effective artificial bone substitutes. It is osteoinductive as well as osteoconductive. These characteristics enable full bone defects regeneration together with its cell-mediated resorption. In this study, we compared between nanocrystalline hydroxyapatite and tricalcium phosphate carried on PRP membrane in treatment of Miller's class 1 gingival recession in human.

ELIGIBILITY:
Inclusion Criteria:

* Patients with good systemic health and no contraindication for periodontal surgery.
* Patients who are able to maintain good oral hygiene.
* Gingival thickness for the site selected should be ≥1mm.
* The height of keratinized gingiva (HKG) for the site selected should be ≥1 mm (HKG is the distance between the most apical point of the gingival margin and the mucogingival junction).

Exclusion Criteria:

* Active infectious diseases (hepatitis, tuberculosis, HIV, etc….).
* Medically compromised patients.
* Patients taking medications known to cause gingival enlargement.
* Pregnant patients and smokers.
* Previous mucogingival surgery at the defect.
* Restorations or caries in the area to be treated and non vital tooth.
* Teeth which are tilted or rotated.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2000-09-01 (Actual); Primary Completion 2022-09-20 (Actual); Study Completion 2023-04-22 (Actual)

PRIMARY OUTCOMES:
Recession height | 6 months
  measurement recession height
Recession width | 6 months
  measurement of Recession width
Height of the keratinized tissue | 6 months
  measurement of Height of the keratinized tissue
Percentage of root coverage | 6 months
  It is calculated after 1, 3, 6 months as [RH preoperative - RH postoperative]/RH preoperative) x 100%.
Radiographic assessment | 6 months
  measurement of buccal bone gain

SECONDARY OUTCOMES:
Probing pocket depth | 6 months
  measurement of Probing pocket depth
Clinical attachment level | 6 months
  measurement of Clinical attachment level

IPD SHARING:
Plan to Share IPD: No